CLINICAL TRIAL: NCT01267760
Title: Clinical and Biochemical Effects of Multipass Hemodialysis
Acronym: MHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Flexdialysis ApS (Unknown)
Responsible Party: Principal Investigator, James heaf, chief physician, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mhd1
Record Dates: First submitted 2010-01-26; First posted 2010-12-28 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Uremia
Keywords: dialysis; hemodialysis; Effect of recycled low-volume dialysate on dialysis efficacy
MeSH Terms: conditions — Uremia | interventions — Dialysis; Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- conventional HD (Active Comparator): conventional 4-hour HD
  Interventions: Device: Multipass hemodialysis

INTERVENTIONS:
Device: Multipass hemodialysis — 8-hour dialysis using a recycled dialysis bath of 25-30 l
  Other Names: dialysis; hemodialysis; dialysate

SUMMARY:
The purpose of this study is to investigate whether recycled dialysis fluid can supply enough clearance for hemodiaysis patients.

DETAILED DESCRIPTION:
Conventional hemodialysis uses large amounts of water, which hinders travel possibilies for home hemodialysis (HD) patients. We have developed a recycling system using 25-30 l dialysate per dialysis. In vitro investigations show that this results in adequate dialysis.

12 HD patients will be studied during two dialysis sessions. The first HD will be a conventional 4 hour dialysis, using single pass dialysate. The second will be an 8-hour HD using multipass (recycled) dialysate 25-30 l. Clearance of urea, creatinine, phosphate and cobalamin will be measured both in the patient and the dialysate. Patient symptoms will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic HD patients
* Informed consent

Exclusion Criteria:

* Age <18 years
* Psychiatric disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Urea Kt/V | 9 hours

SECONDARY OUTCOMES:
Creatinine clearance | 9 hours
Patient symptoms | 9 hours

CONTACTS AND LOCATIONS:
Overall Officials: James G Heaf, MD DMSc, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark, Denmark

REFERENCES:
- [Result] Heaf JG, Axelsen M, Pedersen RS. Multipass haemodialysis: a novel dialysis modality. Nephrol Dial Transplant. 2013 May;28(5):1255-64. doi: 10.1093/ndt/gfs484. Epub 2012 Nov 7. PMID 23136214
- [Derived] Eloot S, Van Biesen W, Axelsen M, Glorieux G, Pedersen RS, Heaf JG. Protein-bound solute removal during extended multipass versus standard hemodialysis. BMC Nephrol. 2015 Apr 18;16:57. doi: 10.1186/s12882-015-0056-y. PMID 25896788